CLINICAL TRIAL: NCT07051759
Title: Assessment of Back Rolls and Algorithm of Management
Brief Title: Back Rolls Assessment
Acronym: Back rolls
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hager Montaser Sayed Bedeer (Other)
Responsible Party: Sponsor-Investigator, Hager Montaser Sayed Bedeer, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Back rolls assessment
Record Dates: First submitted 2025-06-22; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Back Rolls Assesment; Back Rolls Management
Keywords: Back rolls management; Back rolls assessment

STUDY DESIGN:
Intervention Model Description: * Based on determining the main outcome variable, the estimated minimum required sample size is 30 cases.
  * Sample size was calculated using G*power software 3.1.9.7., based on the following assumptions:
  * Main outcome is difference in waist chest ratio in patients before and six months after surgery.
  * Based on clinical experience and after reviewing literatures there is a medium difference.
  * Main statistical test is one tailed paired t test to detect the difference between two means.
  * Effect size =0.5
  * Alpha=0.05
  * Power=0.80
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with back rolls who undergo the back contouring surgery (Experimental)
  Interventions: Procedure: Back contouring surgery

INTERVENTIONS:
Procedure: Back contouring surgery — Back rolls are assessed, and the type of surgery is determined according to grade of back rolls.
  Other Names: Back liposuction; Bra line back lift

SUMMARY:
"Back Rolls" are basically fat deposits on the back in the form of rolls. This is a common problem in women, and concerns were encountered by cosmetic surgeons the worldwide. Deep connective tissue in the back attachments to the underlying muscle and/or periosteum divide the fat deposits on the back into multiple visual compartments. Their nomenclature is based on the anatomical area from where they have originated. The skin-fat envelope is held in place by facial attachments that are named the "zones of adherence".

The extent of fat deposits and number of back rolls, as well as skin laxicity, varies from person to person and also from one side to the other. The rolls surely have a zone of adherence inferiorly over which the tissue fold hangs and medially in the midline. Treatment modalities for back rolls depend on the above-mentioned variables and involve three general approaches:

1. Suction-assisted Liposuction along alone or with other modalities of skin tightening as VASER or J-Plasma ;
2. Direct surgical excision of the skin fold as an upper back lift.
3. Non- surgical: Injection lipolysis in association with weight loss. The choice of treatment depends on the specific characteristic of the back roll; hence, a classification to grade the extent of back roll would help in guiding the surgeon to choose the best possible option.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 50 years old.
* Any grad of back rolls

Exclusion Criteria:

* patients outside the selected age range
* Abnormal laboratory tests (in particular, glucose >105 g/dL, hemoglobin <12 g/dL, platelets <150,000)
* significant systemic diseases.
* previous liposuction or other back surgeries.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
improvement in grading of back rolls | six months postoperative
  Grade I: Back rolls that appear when the arms are kept by the side and disappear when the arms are raised.
  Grade II: Back rolls having a single indentation (partial or complete) that reduces when the arm is raised.
  Grade III: Back rolls with two or more skin indentations with skin pinch of more than 2 cm. The skin fold should not be lower than the inferior tethering point.
  Grade IV: Back rolls secondary to massive weight loss that have multiple folds with skin pinch less than 2 cm and skin fold lower than the tethering point, or in patients who have undergone prior surgical treatment.
Compare the improvement of waist-hip ratio | six months postoperative
  The waist-hip ratio (WHR) is a measurement that compares the circumference of your waist to the circumference of your hips. It's calculated by dividing the waist measurement by the hip measurement.
Compare the improvement of waist-chest ratio | six months postoperative
  The waist-chest ratio is a measurement that compares a person's waist circumference to their chest circumference. It's often used as an indicator of body shape and potential health risks associated with fat distribution.

IPD SHARING:
Plan to Share IPD: No
The majority of patients involved in this type of research are unwilling to disclose personal details beyond the scope of the study itself.

REFERENCES:
- [Background] Thomas MK, D'Silva JA, Borole AJ. Injection Lipolysis: A Systematic Review of Literature and Our Experience with a Combination of Phosphatidylcholine and Deoxycholate over a Period of 14 Years in 1269 Patients of Indian and South East Asian Origin. J Cutan Aesthet Surg. 2018 Oct-Dec;11(4):222-228. doi: 10.4103/JCAS.JCAS_117_18. PMID 30886477
- [Result] Hunstad JP, Repta R. Bra-line back lift. Plast Reconstr Surg. 2008 Oct;122(4):1225-1228. doi: 10.1097/PRS.0b013e3181858fa4. No abstract available. PMID 18827659
- [Result] Mowlavi A, Talle A, Berri M, Rashid W. Successful Back Contouring With Elimination of Back Rolls Using Ultrasound-Assisted Liposuction and Helium-Activated Radiofrequency. Aesthet Surg J Open Forum. 2020 Oct 26;2(4):ojaa036. doi: 10.1093/asjof/ojaa036. eCollection 2020 Dec. PMID 33791662
- [Result] Rohrich RJ, Smith PD, Marcantonio DR, Kenkel JM. The zones of adherence: role in minimizing and preventing contour deformities in liposuction. Plast Reconstr Surg. 2001 May;107(6):1562-9. doi: 10.1097/00006534-200105000-00043. PMID 11335837